CLINICAL TRIAL: NCT03238573
Title: The Real-time Optical Diagnosis Value of Optical Enhancement Endoscopy in Colorectal Sessile Serrated Adenomas/Polyps :A Prospective Study
Brief Title: The Real-time Optical Diagnosis Value of Optical Enhancement Endoscopy in Colorectal Sessile Serrated Adenomas/Polyps
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2017SDU-QILU-03
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Colorectal Sessile Serrated Adenomas/Polyps
Keywords: Colorectal Sessile Serrated Adenomas/Polyps optical enhancement endoscopy
MeSH Terms: conditions — Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- optical enhancment endoscopy

SUMMARY:
When a polyp is found, we begin to wash it and observe it with OE mode 1.Then,the endoscopist gives a real-time optical diagnosis and the future surveillance interval.Finally,the polyp will be resected for the biopsy.

DETAILED DESCRIPTION:
When discovering a polyp, the endoscopist uses water to wash it.Then, the endoscopist starts with i-scan 1 (OE mode 1) to observe the polyp closely .Nextly, the endoscopist give a real-time optical diagnosis with the blind of the history of patient. Considering the other polyps, the endoscopist gives a surveillance interval predictions according to the guide made by USMSTF.The confidence of the real-time optical diagnosis is divided into high confidence and low confidence.After the observation, the small and diminutive polyp will be resected and have the blinded pathology.

ELIGIBILITY:
Inclusion Criteria:

1. The high risk for colorectal cancer screening score
2. Patients with colorectal polyps reviewing

Exclusion Criteria:

* 1.Inflammatory bowel disease 2. Polyposis syndrome 3. A history of colorectal cancer or surgical resection 4. Poor bowel preparation5.Not signing the informed consent 6.Severe cardiopulmonary function failure lesions, severe hypertension, cerebrovascular disease, mental disorder and coma, pregnancy, lactation can't taking the colonoscopy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who experience an examination of coloscopy found polyps
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-07-19 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Real-time diagnosis accuracy of optical enhancement in colorectal sessile serrated adenomas/polyps | 2years

SECONDARY OUTCOMES:
Real-time diagnosis accuracy of optical enhancement in colorectal adenomas and hyperplastic polyps | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Li, MD,PhD, Study Director — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology,Qilu Hospital,Shandong University, Jin'an, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Erichsen R, Baron JA, Hamilton-Dutoit SJ, Snover DC, Torlakovic EE, Pedersen L, Froslev T, Vyberg M, Hamilton SR, Sorensen HT. Increased Risk of Colorectal Cancer Development Among Patients With Serrated Polyps. Gastroenterology. 2016 Apr;150(4):895-902.e5. doi: 10.1053/j.gastro.2015.11.046. Epub 2015 Dec 8. PMID 26677986
- [Result] IJspeert JE, Bastiaansen BA, van Leerdam ME, Meijer GA, van Eeden S, Sanduleanu S, Schoon EJ, Bisseling TM, Spaander MC, van Lelyveld N, Bargeman M, Wang J, Dekker E; Dutch Workgroup serrAted polypS & Polyposis (WASP). Development and validation of the WASP classification system for optical diagnosis of adenomas, hyperplastic polyps and sessile serrated adenomas/polyps. Gut. 2016 Jun;65(6):963-70. doi: 10.1136/gutjnl-2014-308411. Epub 2015 Mar 9. PMID 25753029
- [Result] Lieberman DA, Rex DK, Winawer SJ, Giardiello FM, Johnson DA, Levin TR. Guidelines for colonoscopy surveillance after screening and polypectomy: a consensus update by the US Multi-Society Task Force on Colorectal Cancer. Gastroenterology. 2012 Sep;143(3):844-857. doi: 10.1053/j.gastro.2012.06.001. Epub 2012 Jul 3. No abstract available. PMID 22763141